CLINICAL TRIAL: NCT00671437
Title: Determination of Tumor SUV by FDG-PET/CT Before and After Cetuximab in Patients With Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Determine Tumor Response Using Fluorodeoxyglucose (FDG)- Positron Emission Tomography (PET)/Computed Tomography (CT) Before and After Cetuximab in Patients With Head and Neck Cancer
Acronym: SCCHN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-0285 / 201107108
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma, Squamous Cell
Keywords: squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Whole body FDG-PET/CT scan and CT scan of neck and chest (within 28 days of Day 1)
  Cetuximab 400 mg/m2 intravenously (IV) over 2 hours on day 1 and 250 mg/m2 IV over 1 hour on days 8, 15, 22, 29, 36, 43, and 50.
  Whole Body FDG-PET/CT scan and CT scan of neck and chest on Day 57 (prior to cetuximab infusion)
  Cetuximab 250 mg/m2 IV over 1 hour on Day 57
  Cetuximab 250 mg/m2 IV over 1 hour weekly until progressive disease
  Interventions: Procedure: FDG-PET/CT; Drug: Cetuximab

INTERVENTIONS:
Procedure: FDG-PET/CT
Drug: Cetuximab
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to collect data and evaluate how the tumor is broken down in response to standard of care cetuximab treatment by evaluating the FDG-PET/CT scans, toxicity, see how well the FDG-PET/CT scans predict response to treatment and survival.

DETAILED DESCRIPTION:
Primary Endpoint

To compare the SUV (standardized uptake value) at up to three target tumor sites as assessed by FDG-PET/CT of eligible patients at baseline and then after eight weeks of treatment with cetuximab.

Secondary Endpoints

* To determine the overall tumor metabolic response (complete metabolic response, partial metabolic response, stable metabolic disease or progressive metabolic disease [CMR, PMR, SMD, or PMD]) to eight weeks of scheduled weekly doses of cetuximab as assessed by FDG-PET/CT performed at baseline and then after therapy.
* To correlate the overall tumor metabolic response (CMR, PMR, SMD, or PMD) as assessed by FDG-PET/CT with the anatomic tumor response rate (complete response, partial response, stable disease or progressive disease [CR, PR, SD, or PD]) by RECIST criteria as assessed by CT and clinical examination performed after eight weeks of scheduled weekly doses of cetuximab.
* To correlate the overall tumor metabolic response (CMR, PMR, SMD, or PMD) as assessed by FDG-PET/CT and to correlate the overall anatomic tumor response (CR, PR, SD, or PD) by RECIST criteria as assessed by CT and clinical examination obtained at baseline and after eight weeks of treatment with weekly scheduled doses of cetuximab to TTP (time to progression) and OS (overall survival) with cetuximab therapy.
* To determine the overall best anatomic tumor response rate (CR, PR, SD, or PD) to cetuximab given until disease progression as assessed by RECIST criteria using CT and clinical examination.
* To determine the overall disease control rate (CR, PR, and SD) by RECIST criteria as assessed by CT and clinical examination and to determine the TTP and the OS with cetuximab therapy.
* To assess the toxicity profile for standard of care cetuximab given to patients with metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of squamous cell carcinoma of the head and neck (SCCHN).
* Have either locally recurrent, unresectable, previously irradiated SCCHN OR metastatic SCCHN, with at least one measurable tumor lesion (by CT scan) and at least one FDG avid (SUV >/= 3, >/= 1.5 cm) tumor lesion (by PET/CT).
* Age greater than 18 yrs.
* ECOG Performance Status of 0-3
* Signed IRB approved Informed Consent.

Exclusion Criteria:

* Clinical history of severe interstitial lung disease (not COPD)-as defined by prior pulmonary function tests (PFTs) with residual volume, total lung capacity, or corrected diffuse lung capacity for carbon monoxide (DLCO) <30% of predicted. For this study, screening PFT's required only if clinically indicated.
* Prior therapy with an epidermal growth factor receptor (EGFR)-specific monoclonal antibody (MAB) for treatment of metastatic SCCHN. Prior therapy with an EGFR-specific MAB as part of the definitive treatment of non-metastatic SCCHN is acceptable if this occurred more than three months previously. Prior therapy with an EGFR specific TKI will not be an exclusion factor.
* Women of child bearing potential who are current pregnant or breast feeding.
* Prior severe (Grade 4) infusion reaction to cetuximab.
* A serious uncontrolled medical disorder that in the opinion of the Investigator would impair the ability of the subject to receive protocol therapy.
* Chemotherapy, radiation therapy, or investigational agents given with the last 14 days.
* Uncontrolled diabetes mellitus. (Subjects with a fasting blood glucose > 200 at time of PET scanning may need to reschedule to another day after consulting with appropriate physicians.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Louisville, Louisville, Kentucky
  - Washington University, St Louis, Missouri

REFERENCES:
- [Background] Jemal A, Tiwari RC, Murray T, Ghafoor A, Samuels A, Ward E, Feuer EJ, Thun MJ; American Cancer Society. Cancer statistics, 2004. CA Cancer J Clin. 2004 Jan-Feb;54(1):8-29. doi: 10.3322/canjclin.54.1.8. PMID 14974761
- [Background] Mendelsohn J, Baselga J. Status of epidermal growth factor receptor antagonists in the biology and treatment of cancer. J Clin Oncol. 2003 Jul 15;21(14):2787-99. doi: 10.1200/JCO.2003.01.504. PMID 12860957
- [Background] Dassonville O, Formento JL, Francoual M, Ramaioli A, Santini J, Schneider M, Demard F, Milano G. Expression of epidermal growth factor receptor and survival in upper aerodigestive tract cancer. J Clin Oncol. 1993 Oct;11(10):1873-8. doi: 10.1200/JCO.1993.11.10.1873. PMID 8410112
- [Background] Ang KK, Berkey BA, Tu X, Zhang HZ, Katz R, Hammond EH, Fu KK, Milas L. Impact of epidermal growth factor receptor expression on survival and pattern of relapse in patients with advanced head and neck carcinoma. Cancer Res. 2002 Dec 15;62(24):7350-6. PMID 12499279
- [Background] Huang S, Armstrong EA, Benavente S, Chinnaiyan P, Harari PM. Dual-agent molecular targeting of the epidermal growth factor receptor (EGFR): combining anti-EGFR antibody with tyrosine kinase inhibitor. Cancer Res. 2004 Aug 1;64(15):5355-62. doi: 10.1158/0008-5472.CAN-04-0562. PMID 15289342
- [Background] Cohen EE, Rosen F, Stadler WM, Recant W, Stenson K, Huo D, Vokes EE. Phase II trial of ZD1839 in recurrent or metastatic squamous cell carcinoma of the head and neck. J Clin Oncol. 2003 May 15;21(10):1980-7. doi: 10.1200/JCO.2003.10.051. PMID 12743152
- [Background] Bonner JA, Harari PM, Giralt J, Azarnia N, Shin DM, Cohen RB, Jones CU, Sur R, Raben D, Jassem J, Ove R, Kies MS, Baselga J, Youssoufian H, Amellal N, Rowinsky EK, Ang KK. Radiotherapy plus cetuximab for squamous-cell carcinoma of the head and neck. N Engl J Med. 2006 Feb 9;354(6):567-78. doi: 10.1056/NEJMoa053422. PMID 16467544
- [Background] Baselga J, Trigo JM, Bourhis J, Tortochaux J, Cortes-Funes H, Hitt R, Gascon P, Amellal N, Harstrick A, Eckardt A. Phase II multicenter study of the antiepidermal growth factor receptor monoclonal antibody cetuximab in combination with platinum-based chemotherapy in patients with platinum-refractory metastatic and/or recurrent squamous cell carcinoma of the head and neck. J Clin Oncol. 2005 Aug 20;23(24):5568-77. doi: 10.1200/JCO.2005.07.119. Epub 2005 Jul 11. PMID 16009950
- [Background] J. Trigo et al., Cetuximab monotherapy is active in patients with platinum-refractory recurrent/metastatic squamous cell carcinoma of the head and neck: Results of a phase II study (abstract). Proc Am Soc Clin Oncol 23 (2004), p. 487a.
- [Background] Vermeersch H, Loose D, Ham H, Otte A, Van de Wiele C. Nuclear medicine imaging for the assessment of primary and recurrent head and neck carcinoma using routinely available tracers. Eur J Nucl Med Mol Imaging. 2003 Dec;30(12):1689-700. doi: 10.1007/s00259-003-1345-4. Epub 2003 Oct 22. PMID 14574516
- [Background] Antoch G, Saoudi N, Kuehl H, Dahmen G, Mueller SP, Beyer T, Bockisch A, Debatin JF, Freudenberg LS. Accuracy of whole-body dual-modality fluorine-18-2-fluoro-2-deoxy-D-glucose positron emission tomography and computed tomography (FDG-PET/CT) for tumor staging in solid tumors: comparison with CT and PET. J Clin Oncol. 2004 Nov 1;22(21):4357-68. doi: 10.1200/JCO.2004.08.120. PMID 15514377
- [Background] Schwartz DL, Rajendran J, Yueh B, Coltrera MD, Leblanc M, Eary J, Krohn K. FDG-PET prediction of head and neck squamous cell cancer outcomes. Arch Otolaryngol Head Neck Surg. 2004 Dec;130(12):1361-7. doi: 10.1001/archotol.130.12.1361. PMID 15611393
- [Background] Minn H, Lapela M, Klemi PJ, Grenman R, Leskinen S, Lindholm P, Bergman J, Eronen E, Haaparanta M, Joensuu H. Prediction of survival with fluorine-18-fluoro-deoxyglucose and PET in head and neck cancer. J Nucl Med. 1997 Dec;38(12):1907-11. PMID 9430467
- [Background] Brun E, Kjellen E, Tennvall J, Ohlsson T, Sandell A, Perfekt R, Perfekt R, Wennerberg J, Strand SE. FDG PET studies during treatment: prediction of therapy outcome in head and neck squamous cell carcinoma. Head Neck. 2002 Feb;24(2):127-35. doi: 10.1002/hed.10037. PMID 11891942
- [Background] Weber WA, Ott K, Becker K, Dittler HJ, Helmberger H, Avril NE, Meisetschlager G, Busch R, Siewert JR, Schwaiger M, Fink U. Prediction of response to preoperative chemotherapy in adenocarcinomas of the esophagogastric junction by metabolic imaging. J Clin Oncol. 2001 Jun 15;19(12):3058-65. doi: 10.1200/JCO.2001.19.12.3058. PMID 11408502
- [Background] Choi NC, Fischman AJ, Niemierko A, Ryu JS, Lynch T, Wain J, Wright C, Fidias P, Mathisen D. Dose-response relationship between probability of pathologic tumor control and glucose metabolic rate measured with FDG PET after preoperative chemoradiotherapy in locally advanced non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2002 Nov 15;54(4):1024-35. doi: 10.1016/s0360-3016(02)03038-9. PMID 12419428
- [Background] Kostakoglu L, Coleman M, Leonard JP, Kuji I, Zoe H, Goldsmith SJ. PET predicts prognosis after 1 cycle of chemotherapy in aggressive lymphoma and Hodgkin's disease. J Nucl Med. 2002 Aug;43(8):1018-27. PMID 12163626
- [Background] M. Beeram et al., Durable disease stabilization and antitumor activity with OSI-774 in renal cell carcinoma: A phase II, pharmacokinetic (PK) and biological correlative study with FDG-PET imaging. J Clinical Oncology 22 (2004), pp. 3050.
- [Background] T. Trarbach et al., A randomized phase I study of the humanized anti-epidermal growth factor receptor (EGFR) monoclonal antibody EMD 72000 in subjects with advanced gastrointestinal cancers. J Clinical Oncology 22 (2004), pp. 3018.
- [Background] Goldstein D, Tan BS, Rossleigh M, Haindl W, Walker B, Dixon J. Gastrointestinal stromal tumours: correlation of F-FDG gamma camera-based coincidence positron emission tomography with CT for the assessment of treatment response--an AGITG study. Oncology. 2005;69(4):326-32. doi: 10.1159/000089765. Epub 2005 Nov 16. PMID 16293972
- [Background] Antoch G, Kanja J, Bauer S, Kuehl H, Renzing-Koehler K, Schuette J, Bockisch A, Debatin JF, Freudenberg LS. Comparison of PET, CT, and dual-modality PET/CT imaging for monitoring of imatinib (STI571) therapy in patients with gastrointestinal stromal tumors. J Nucl Med. 2004 Mar;45(3):357-65. PMID 15001674
- [Background] Gayed I, Vu T, Iyer R, Johnson M, Macapinlac H, Swanston N, Podoloff D. The role of 18F-FDG PET in staging and early prediction of response to therapy of recurrent gastrointestinal stromal tumors. J Nucl Med. 2004 Jan;45(1):17-21. PMID 14734662
- [Background] Bristol-Meyer-Squibb, Product Information for Erbitux, 2004.
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was open from 06/03/08-10/17/11 at the Siteman Cancer Center (a medical clinic).
Groups:
- Arm 1 (Cetuximab): Whole body Fluorodeoxyglucose (FDG)- Positron Emission Tomography (PET)/Computed Tomography (CT) scan and CT scan of neck and chest (within 28 days of Day 1)
  Cetuximab 400 mg/m2 intravenously (IV) over 2 hours on day 1 and 250 mg/m2 IV over 1 hour on days 8, 15, 22, 29, 36, 43, and 50.
  Whole Body FDG-PET/CT scan and CT scan of neck and chest on Day 57 (prior to cetuximab infusion)
  Cetuximab 250 mg/m2 IV over 1 hour on Day 57
  Cetuximab 250 mg/m2 IV over 1 hour weekly until progressive disease
Period: Overall Study
Arm/Group | Arm 1 (Cetuximab)
Started | 42
Completed | 27
Not Completed | 15
Not completed — Progressive disease before C1 week 8 | 8
Not completed — Cutaneous SCC of head and neck | 3
Not completed — Adverse Event | 3
Not completed — Ineligible post-hoc | 1

BASELINE CHARACTERISTICS:
Population: Baseline participants are based on the number of evaluable patients. 15 out of the 42 enrolled patients were not considered evaluable for analyses.
Groups:
- Arm 1 (Cetuximab): Whole body FDG-PET/CT scan and CT scan of neck and chest (within 28 days of Day 1)
  Cetuximab 400 mg/m2 IV over 2 hours on day 1 and 250 mg/m2 IV over 1 hour on days 8, 15, 22, 29, 36, 43, and 50.
  Whole Body FDG-PET/CT scan and CT scan of neck and chest on Day 57 (prior to cetuximab infusion)
  Cetuximab 250 mg/m2 IV over 1 hour on Day 57
  Cetuximab 250 mg/m2 IV over 1 hour weekly until progressive disease
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 63 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status Grade 0 Fully active able to carry on all predisease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (light house work/office work)
  2. Ambulatory, capable of all selfcare but unable to carry out any work activities. Up & about more than 50% of waking hours
  3. Capable of limited selfcare, confined to bed/chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on selfcare. Totally confined to bed/chair
  5. Dead
  participants
    Performance Status 0 | 5
    Performance Status 1 | 13
    Performance Status 2 | 9
Smoking history [Number; unit: participants]
  Yes | 24
  No | 3
Primary Tumor Site [Number; unit: participants]
  Oral cavity | 10
  Oropharynx | 8
  Larynx | 4
  Hypopharynx | 5
Prior Cetuximab Exposure [Number; unit: participants]
  Yes | 8
  No | 19

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Response of Target Lesions Assessed as the Change in Standardized Uptake Values (SUV) Max on FDG-PET/CT
Description: FDG-PET/CT images were evaluated qualitatively as well as quantitatively by one of two experienced nuclear radiologists. For quantitative analysis, SUVmax within each of the metastatic tumor sites was determined within a volume of interest around the tumor using a Siemens eSoft workstation. Up to a maximum of three target lesions(>= 1.5 cm on the baseline CT) were identified as target lesions on the baseline FDG-PET. When multiple lesions were present, those having the greatest FDG uptake on the baseline FDG-PET were selected as target lesions. Lesions containing areas of necrosis were avoided. Other metabolically active lesions and lesions that were <1.5 cm on CT were considered non-target lesions. When more than one target lesion was identified, the average percentage change in SUVmax was used to determine metabolic response.
Time Frame: Baseline and after 8 weeks of treatment
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 27
percentage of change | -21 [-81 to 72]

2. Primary Outcome: SUVmax at up to Three Target Tumor Sites as Assessed by FDG-PET/CT of Eligible Patients at Baseline and Then After Eight Weeks of Treatment With Cetuximab.
Description: Eight weeks of treatment is equal to one cycle of treatment.
  FDG-PET/CT images were evaluated qualitatively as well as quantitatively by one of two experienced nuclear radiologists. For quantitative analysis, SUVmax within each of the metastatic tumor sites was determined within a volume of interest around the tumor using a Siemens eSoft workstation. Up to a maximum of three target lesions(>= 1.5 cm on the baseline CT) were identified as target lesions on the baseline FDG-PET. When multiple lesions were present, those having the greatest FDG uptake on the baseline FDG-PET were selected as target lesions. Lesions containing areas of necrosis were avoided. Other metabolically active lesions and lesions that were <1.5 cm on CT were considered non-target lesions. When more than one target lesion was identified, the average percentage change in SUVmax was used to determine metabolic response.
Time Frame: Baseline and after 8 weeks of treatment
Measure: Mean (95% Confidence Interval); unit: SUVmax
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 27
SUVmax
  Pre-Cetuximab | 9.3 [7.2 to 12.1]
  Post Cycle 1 | 7.3 [5.6 to 9.5]

3. Secondary Outcome: Overall Tumor Metabolic Response to Eight Weeks of Scheduled Weekly Doses of Cetuximab as Assessed by FDG-PET/CT
Description: Definitions of metabolic response by FDG-PET/CT included: complete metabolic response(CMR)-complete resolution of all metabolically active target and non-target lesions, and no new lesions; partial metabolic response(PMR)-20% or greater decrease in SUV of target lesions with or without decrease in number/size of non-target lesions, and no new lesions; progressive metabolic disease(PMD)-one or more new lesions, 20% or greater increase in SUV of target lesions and/or unequivocal increase in FDG activity of non-target lesions; and stable metabolic disease(SMD)-not qualifying as CMR, PMR, or PMD.
Time Frame: After 8 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 27
participants
  PMR/SMD | 15
  PMD | 12

4. Secondary Outcome: Overall Anatomic Response to Eight Weeks of Scheduled Weekly Doses of Cetuximab as Assessed by CT Scan
Description: Definitions of anatomic response by RECIST for CT scan included: complete response(CR)-disappearance of all target and non-target lesions and no new lesions; partial response(PR)-at least 30% decrease in the sum of the longest diameter of target lesions taking as reference the baseline sum longest diameter, persistence of one or more non-target lesions, and no new lesions; stable disease (SD)-neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum longest diameter since the treatment started, persistence of one or more non-target lesions, and no new lesions; progressive disease(PD)-at least a 20% increase in the sum of the longest diameter of target lesions recorded since the treatment started, appearance of one or more new lesions/unequivocal progression of existing non-target lesions.
Time Frame: After 8 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 27
participants
  Partial Response/Stable Disease | 20
  Progressive Disease | 7

5. Secondary Outcome: Correlation of Overall Tumor Metabolic Response as Assessed by FDG-PET/CT With the Anatomic Tumor Response Rate by RECIST Criteria as Assessed by CT and Clinical Examination
Description: A generalization of McNemar's test was used to test for concordance of response(partial, stable or progression) by CT and by FDG-PET/CT.
Time Frame: After 8 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Partial Metabolic Response (Overall PET Response) | Stable Metabolic Disease (Overall PET Response) | Progressive Metabolic Disease (Overall PET Response) | Total (Overall PET Response)
Number analyzed (Participants) | 10 | 5 | 12 | 27
participants
  Partial Response (overall CT response) | 1 | 0 | 0 | 1
  Stable Disease (overall CT response) | 9 | 5 | 5 | 19
  Progressive Disease (overall CT response) | 0 | 0 | 7 | 7
  Total (overall CT response) | 10 | 5 | 12 | 27

6. Secondary Outcome: Correlation of Overall Tumor Metabolic Response as Assessed by FDG-PET/CT With the Anatomic Tumor Response Rate by RECIST Criteria as Assessed by CT and Clinical Examination
Description: Agreement in treatment decision using CT and FDG-PET/CT. Agreement in treatment decision occurred when tumor response by CT and FDG-PET/CT resulted in the same decision in treatment (continue cetuximab due to disease control or stop cetuximab due to progression). Disagreement in treatment decision occurred when tumor response assessment by CT and FDG-PET/CT resulted in different treatment decisions.
Time Frame: After 8 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 27
participants
  Treatment Agreement | 22
  Treatment Disagreement | 5

7. Secondary Outcome: Overall Best Anatomic Tumor Response Rate to Cetuximab Given Until Disease Progression as Assessed by RECIST Criteria Using CT & Clinical Examination
Time Frame: Every 8 weeks until disease progression (up to 1 year)
Measure: Number; unit: participants
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 27
participants
  Partial Response | 1
  Stable Disease | 20
  Progressive Disease | 7

8. Secondary Outcome: Correlate the Overall Tumor Metabolic Response and Overall Anatomic Tumor Response and Clinical Examination Obtained at Baseline and After Eight Weeks of Treatment With Cetuximab to Time to Progression (TTP) With Cetuximab Therapy
Description: Cetuximab was continued after cycle 1 in patients with disease control(PR/SD) by CT, even if the FDG-PET/CT showed PMD. Cetuximab was discontinued after cycle 1 in patients with progression by CT.
Time Frame: Every 8 weeks until disease progression (up to 1 year)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Disease Control by CT and PET/CT | Disease Control by CT and Progressive Disease by PET/CT | Progressive Disease by Both CT and PET/CT
Number analyzed (Participants) | 15 | 5 | 7
days | 166 [86 to 217] | 105 [66 to 159] | 53 [49 to 56]

9. Secondary Outcome: Correlate the Overall Tumor Metabolic Response and Overall Anatomic Tumor Response and Clinical Examination Obtained at Baseline and After Eight Weeks of Treatment With Cetuximab to Overall Survival With Cetuximab Therapy
Time Frame: Every 8 weeks until death (approximately 5 years)
Population: The small dataset precluded an adequate analysis of overall survival relationships due to varying co-variates such as post-progression therapies, ECOG PS, co-morbidities.
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 0

10. Secondary Outcome: Determine the Overall Disease Control Rate by RECIST Criteria as Assessed by CT and Clinical Examination and to Determine the TTP and the OS With Cetuximab Therapy
Time Frame: Every 8 weeks until death (approximately 5 years)
Population: This was not analyzed due to the lack of evidence-based medicine showing an overall survival benefit of cetuximab monotherapy in this type of cancer.
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 0

11. Secondary Outcome: Assess the Toxicity Profile for Standard of Care Cetuximab Given to Patients With Metastatic Squamous Cell Carcinoma of the Head and Neck
Time Frame: 30 days after end of study treatment (approximately 1 year after start of treatment)
Measure: Number; unit: participants
Arm/Group | Arm 1 (Cetuximab)
Number analyzed (Participants) | 27
participants
  Allergic reaction/hypersensitivity | 5
  Hypotension | 1
  INR | 9
  PTT | 8
  Fever | 1
  Fatigue | 15
  Insomnia | 1
  Rigors | 1
  Weight loss | 7
  Failure to thrive | 1
  Death - progression | 1
  Alopecia | 1
  Bruising - port site | 1
  Bruising - thigh | 1
  Rash/desquamation | 3
  Chelitis | 1
  Dry skin | 7
  Rash - acneiform | 28
  Rash - trach site | 1
  Anorexia | 3
  Constipation | 7
  Dehydration | 2
  Diarrhea | 5
  Dry mouth | 1
  Dysphagia | 1
  Mucositis | 4
  Nausea | 13
  Taste alteration | 1
  Vomiting | 2
  Hemoglobin | 21
  Leukopenia | 3
  Lymphopenia | 27
  Platelets | 2
  Hemorrhage: nose | 1
  Hemorrhage: oral cavity | 1
  Hemorrhage: pulmonary | 1
  Hemorrhage: tumor site | 3
  Alkaline phosphatase | 6
  Bilirubin | 3
  SGOT (AST) | 6
  SGPT (ALT) | 9
  Infection without neutropenia | 1
  Infection normal ANC - cellulitis | 2
  Infection normal ANC - left neck wound | 1
  Infection normal ANC - sinus | 1
  Infection normal ANC - scalp drainage Ecoli | 1
  Infection normal ANC - scalp wound | 1
  Infection normal ANC - skin | 3
  Infection normal ANC - staph shingles | 1
  Infection normal ANC - tumor | 1
  Infection normal ANC - upper respiratory | 2
  Infection normal ANC - urinary tract infection | 1
  Infection normal ANC - yeast | 1
  Infection lung - pneumonia | 2
  Infection skin - ungual | 9
  Edema - eye | 1
  Edema - head & neck | 2
  Edema - limb | 4
  Albumin - low | 26
  Calcium - low | 18
  Calcium - high | 2
  Glucose - low | 3
  Glucose - high | 9
  Magnesium - low | 14
  Magnesium - high | 2
  Phosphorus - low | 3
  Potassium - low | 8
  Potassium - high | 5
  Sodium - low | 14
  Sodium - high | 5
  Fracture | 1
  Brachial plexophathy | 1
  Mood alteration - anxiety | 1
  Mood alteration - depression | 1
  Restless leg | 1
  Syncope | 1
  Back pain | 2
  Headache | 2
  Neck pain | 3
  Tumor pain | 5
  Aspiration | 1
  Bronchospasm/wheezing | 1
  Cough | 2
  Dyspnea | 4
  Hypoxia | 2
  Voice changes/dysarthria | 1
  Creatinine | 9
  Diuresis | 1
  Dry eye syndrome | 1
  Thrombosis | 1
  Trismus | 1

ADVERSE EVENTS:
Arm/Group | Arm 1 (Cetuximab)
Serious Adverse Events (participants affected / at risk) | 7/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Cetuximab) (N=42)
Allergic reaction/hypersensitivity (Immune system disorders) | 1 (1) — Grade 4
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1) — Grade 4
Brachial plexopathy (Nervous system disorders) | 1 (1) — Grade 4 Due to radiographically proven tumor progression
Bronchospasm/Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 5 Chronic obstructive pulmonary disease (COPD)
Death - Disease Progression (General disorders) | 1 (1) — Grade 5
Infection lung - pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 5
Lymphocytes (decreased) (Investigations) | 1 (1) — Grade 4 Occurred in the setting of concurrent administration of dexamethasone for head and neck lymph edema occurring due to the patient's disease.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Cetuximab) (N=42)
Albumin (low) (Metabolism and nutrition disorders) | 26
Alkaline phosphatase (high) (Investigations) | 6
Allergic reaction/hypersensitivity (Immune system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 3
Bilirubin (hyperbilirubinemia) (Investigations) | 2
Calcium (high) (Metabolism and nutrition disorders) | 2
Calcium (low) (Metabolism and nutrition disorders) | 18
Constipation (Gastrointestinal disorders) | 7
Creatinine (high) (Investigations) | 9
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 7
Edema - head and neck (General disorders) | 2
Edema - limb (General disorders) | 4
Fatigue (General disorders) | 15
Glucose (high) (Metabolism and nutrition disorders) | 9
Glucose (low) (Metabolism and nutrition disorders) | 3
Headache (Nervous system disorders) | 2
Hemoglobin (low) (Blood and lymphatic system disorders) | 21
Hemorrhage: Tumor Site (Vascular disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
INR (high) (Investigations) | 9
Infection normal ANC - cellulitis (Infections and infestations) | 2
Infection normal ANC - skin (Infections and infestations) | 3
Infection normal ANC - upper respiratory (Infections and infestations) | 2
Infection skin - ungual (Infections and infestations) | 9
Leukocytes (low) (Investigations) | 3
Lymphocytes (low) (Investigations) | 26
Magnesium (high) (Metabolism and nutrition disorders) | 2
Magnesium (low) (Metabolism and nutrition disorders) | 14
Mucositis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 13
PTT (high) (Investigations) | 8
Pain - back (Musculoskeletal and connective tissue disorders) | 2
Pain - musculoskeletal - neck (Musculoskeletal and connective tissue disorders) | 3
Phosphate (low) (Metabolism and nutrition disorders) | 3
Platelets (low) (Investigations) | 2
Potassium (low) (Metabolism and nutrition disorders) | 8
Rach - acneiform (Skin and subcutaneous tissue disorders) | 28
Rash - trach site (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
SGOT (AST - high) (Investigations) | 6
SGPT (ALT-high) (Investigations) | 9
Sodium (high) (Metabolism and nutrition disorders) | 5
Sodium (low) (Metabolism and nutrition disorders) | 14
Vomiting (Gastrointestinal disorders) | 2
Weight loss (Investigations) | 7
Potassium (high) (Metabolism and nutrition disorders) | 5
Pain - tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No